CLINICAL TRIAL: NCT05664659
Title: Carbetocin Versus Oxytocin Plus Misoprostol in Decreasing Intraoperative Blood Loss in Women Undergoing Planned Cesarean Section
Brief Title: Efficacy of Carbetocin Versus Oxytocin Plus Misoprostol in Decreasing Blood Loss During Cesarean Section
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams Maternity Hospital (Other)
Responsible Party: Principal Investigator, Rania Hassan Mostafa, Principal investigator, Ain Shams Maternity Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: FMASU MS 211/2022
Record Dates: First submitted 2022-12-16; First posted 2022-12-27 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Blood Loss, Surgical; Intrapartum Hemorrhage
Keywords: estimated blood loss; carbetocin; oxytocin; misoprostol
MeSH Terms: conditions — Blood Loss, Surgical | interventions — Oxytocin; Misoprostol; carbetocin

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Eligible patients will be randomised & allocated into 2 groups (A) & (B). Randomization will be done using computer generated list.
  Allocation & concealment will be done using sealed envelopes prepared according to computer generated list into ratio 1:1.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oxytocin+Misoprostol (Active Comparator): Patients in this group will receive 600 micrograms misoprostol rectally immediately before sterilization plus 20 IU Oxytocin IV infusion on 1000 ml of normal saline solution immediately after delivery of the fetus.
  Interventions: Drug: Oxytocin + misoprostol
- Carbetocin (Experimental): Patients in this group will receive 100ug Carbetocin by slow IV infusion (over one minute) intra-operative immediately after delivery of the fetus.
  Interventions: Drug: Carbetocin

INTERVENTIONS:
Drug: Oxytocin + misoprostol — 600 micrograms misoprostol rectally 20 IU Oxytocin IV infusion on 1000 ml of normal saline solution
  Arms: Oxytocin+Misoprostol
Drug: Carbetocin — 100 micrograms carbetocin
  Arms: Carbetocin

SUMMARY:
The aim of this clinical trial is to test if carbetocin is as effective as oxytocin plus misoprostol in decreasing intraoperative blood loss in women undergoing planned cesarean section.

The main question it aims to answer is:

* Is carbetocin as effective as oxytocin plus misoprostol in decreasing intraoperative blood loss in women undergoing planned cesarean section?

Researchers will compare 2 groups:

* women receiving Oxytocin plus Misoprostol;
* women receiving Carbetocin as regards:
* estimated blood loss

DETAILED DESCRIPTION:
* Type of Study: A randomized controlled clinical trial.
* Study Setting: This study will be conducted in Ain Shams University Maternity Hospital (ASUMH).
* Study duration: 6 months.
* Study population: Women will be recruited from outpatient antenatal clinic of ASUMH.

Sample Size:

104 patients will be enrolled in this study and will be divided into two groups:

* Group A: 52 patients will receive+ Oxytocin (20 IU IV infusion on 1000 ml of normal saline solution) plus misoprostol (600 micrograms rectal). ( The control group )
* Group B: 52 patients will receive 100 micrograms Carbetocin IV slowly. Sample size justification By using PASS 11 software for sample size calculation, setting power at 80%, alpha error at 5% and after reviewing previous study results showed that the haemoglobin level (g/dl) postoperative to caesarean section was higher among women took Carbetocin than those took misoprostol (10.13 ± 0.76 versus 9.57 ± 0.95 respectively); based on that, a sample size of at least 90 pregnant females undergoing elective caesarean section divided randomly into 2 intervention groups [Carbetocin and misoprostol with oxytocin] (45 patients in each group) will be sufficient to achieve study objective, yet the drop out rate 17% so 7 patients will be added in each group.

Procedures:

1. Approval of the protocol by the ethical committee of the department of Obstetrics & Gynecology, Faculty of Medicine, Ain Shams University.
2. Recruitment of patients planning to undergo elective cesarean section in ASUMH from antenatal clinic.
3. An informed written consent will be taken from all participants before enrollment in the study and after explaining the purpose, possible risks and complications.
4. All participants will be subjected to thorough history taking, general and abdominal examination, obstetric ultrasound examination and laboratory investigations including complete blood count to identify eligible patients.
5. The expert consultant will take the decision to do the cesarean section.
6. Eligible patients will be randomised & allocated into 2 groups (A) & (B). Randomization will be done using computer generated list.
7. Allocation & concealment will be done using sealed envelopes prepared according to computer generated list into ratio 1:1. Patients will deliver by cesarean section. Patients in group A will receive 600 micrograms misoprostol rectally immediately before sterilization plus 20 IU Oxytocin IV infusion on 1000 ml of normal saline solution immediately after delivery of the fetus.
8. Patients in group B will receive 100ug Carbetocin by slow IV infusion (over one minute) intra-operative immediately after delivery of the fetus.
9. Estimation of blood loss will be calculated by :

   * After delivery of the placenta, the amount of blood loss in the suction canister and drapes will be measured.
   * The equation* used when calculating blood loss of a blood-soaked item is WET Item Gram Weight - DRY Item Gram Weight=Milliliters of Blood Within the Item. The items are weighed using a highly accurate digital balance ( Salter digital electronic scale 9037 TL3R).
   * Although a gram is a unit of mass and a milliliter is a unit of volume, the conversion from one to the other is a simple 1-to-1 conversion.
   * The amniotic fluid index (AFI) was estimated using abdominal ultrasound as the sum of the maximum vertical diameter of amniotic fluid in four quadrants in centimeters.
   * Amniotic fluid volume (AFV) (ml) was estimated by multiplying AFI (cm) by 30.
   * At the end of the surgery, the volume of quantified blood calculated by weight will be added to the volume of quantified blood in the suction canister then subtracting the amniotic fluid volume to determine total quantification of blood loss.
10. Follow up & data recording; • Post-partum hemorrhage will be considered:

1. Minor PPH: if estimated blood loss from 500 ml to 1000 ml. 2. Major PPH: if any estimated blood loss is more than 1000 ml.

* Measuring hemoglobin level before & after 24 hours of delivery to asses the need for blood transfusion.
* All data will be recorded in Case Report Form.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women planning to deliver by CS.
* Age between 18-40.
* Gestational age: (36-42 weeks).

Exclusion Criteria:

1. Women in active labour.
2. Rupture of membranes more than 24 hours &/or intraamniotic infection.
3. Suspected extensive adhesions eg: more than P3CS, endometriosis, previous pelvic surgery.
4. Antepartum hemorrhage and abnormal placentation e.g.: low lying placenta, placenta previa, placenta accreta.
5. Major intrapartum hemorrhage more than 1000 ml.
6. History of postpartum hemorrhage.
7. Anemia (Hb level less than 10g/dl).
8. Uterine overdistention eg: polyhydramnios, macrosomic baby, multiple pregnancy.
9. Known allergy to any of misoprostol, oxytocin, carbetocin.
10. Known medical disorders: Diabetes Mellitus, hypertensive disorders, Systemic Lupus Erythematosus.
11. Known coagulopathy problem.
12. Contraindication &/or refusal to spinal anesthesia.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2022-12-20 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-05-20 (Actual)

PRIMARY OUTCOMES:
estimated blood loss in millimeters | calculated once at the end of the CS
  estimated blood lost during the cesarean section (CS)

SECONDARY OUTCOMES:
drop in hemoglobin | calculated once after 24hours of the CS
  Difference in Hemoglobin level before and after CS

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed SE Sweed, MD, Study Director — Ain Shams University
Locations (1):
- Ain Shams Maternity Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The study protocol and the analytic code will be made available from the central contact on reasonable requests
Supporting Information: Study Protocol, Analytic Code
Time Frame: Data will be available after completion of the study and publishing the results, for 5 years therafter.
Access Criteria: requests for data are to be sent at: raneyah@gmail.com